CLINICAL TRIAL: NCT06683794
Title: The Prognostic Value of the AST/ALT Ratio Vs. APACHE II Score in Patients with Sepsis and Septic Shock
Brief Title: Predicts Mortality by AST/ALT Ration in Patients with Sepsis and Septic Shock During ICU Admissin
Status: Not yet recruiting | Type: Observational
Sponsor: Nermeen Gamil Ahmed (Other)
Responsible Party: Sponsor-Investigator, Nermeen Gamil Ahmed, resident doctors at internal medicine department, Assiut University
Organization: Assiut University (Other)
Other Study IDs: AST/ALT VS APACHE II in Predic
Record Dates: First submitted 2024-10-20; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: E Prognostic Value of the AST/ALT Ratio Vs. APACHE II Score in Patients with Sepsis and Septic Shock
Keywords: AST/ALT ratio
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
1_The study predicts mortality by using Asparate aminotransferase (AST) to Alanine aminotransferase (ALT) ratio in patients with sepsis and septic shock during the duration of ICU admission and for one month after discharge.

2- Compare between APACHE II and AST/ALT ratio as prognostic factors in patients with sepsis and septic shock.

DETAILED DESCRIPTION:
Sepsis is characterized by dysregulated host responses to an infection and may lead to life-threatening organ dysfunctions. Despite recent improvements in the therapy of sepsis including early-goal-directed therapy and improved adherence to treatment guidelines, sepsis is still associated with significant morbidity and mortality. Clinical evidence has shown that hepatic dysfunction is an early event in sepsis, and is an independent risk factor for poor outcome. Clinical manifestations of sepsis-associated liver dysfunction include hypoxic hepatitis, sepsis-induced cholestasis and dysfunction of protein synthesis manifesting with, e.g., coagulopathies . Aspartate aminotransferase (AST) is present in both the cytoplasm and mitochondria of tissue cells, such as the liver, skeletal muscle, heart, brain, and even the kidney, whereas alanine transaminase (ALT) is predominantly located in the cytoplasm of liver tissue. It is thought that ALT primarily reflects liver-specific malfunction, whereas AST may indicate mitochondrial dysfunction resulting from oxidative stress in other tissues to a certain degree. Increases in the AST/ALT ratio indicates systemic derangements such as increased oxidative stress, inflammatory response, and ischemic-reperfusion injury , but might also play a role in more systemic derangements such as increased oxidative stress, inflammatory response, and ischemic-reperfusion injury Limited data regarding the prognostic value of the AST/ALT ratio in patients suffering from sepsis or septic shock is available . The APACHE II (Acute Physiology and Chronic Health Evaluation II) score is a severity-of-disease classification system used to assess the prognosis of critically ill patients. It was developed to predict the risk of hospital mortality and is commonly used in intensive care units (ICUs) to evaluate the severity of illness in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients admitted to the ICU with a diagnosis of sepsis or septic shock according to the Surviving Sepsis Campaign criteria. Diagnostic Criteria for Sepsis and Septic Shock (Sepsis-3) Sepsis: Life-threatening organ dysfunction caused by a dysregulated host response to infection. Organ dysfunction is identified as an acute change in total SOFA (Sequential organ failure assessment) score ≥2 points due to infection.

Septic Shock: A subset of sepsis where underlying circulatory and cellular/metabolic abnormalities are profound enough to substantially increase mortality. Patients with septic shock can be clinically identified by a vasopressor requirement to maintain a mean arterial pressure (MAP) of 65 mm Hg or greater and a serum lactate level >2 mmol/L in the absence of hypovolemia.

Exclusion Criteria:Patients with pre-existing liver disease e.g. chronic hepatitis or cirrhosis.

2. Patients with a history of alcohol abuse. 3. Patients on high dose statin therapy. 4. patients with other causes that could raise AST and ALT e,g, rhabdomyolysis, myocardial infarction.

4. Patients with missed data or who couldnt be followed up

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients admitted to the ICU with a diagnosis of sepsis or septic shock according to the Surviving Sepsis Campaign criteria. Diagnostic Criteria for Sepsis and Septic Shock (Sepsis-3)
Sampling Method: Non-Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The accuracy of the AST/ALT ratio as prognostic factors in patients with sepsis and septic shock | During duration of ICU admission and for 1 month after discharge
  The accuracy of using Asparate aminotransferase (AST) to Alanine aminotransferase (ALT) ratio in patients with sepsis and septic shock to predict mortality during the duration of ICU admission and for one month after discharge.

SECONDARY OUTCOMES:
sensitivity of AST/ALT ratio compare to APACHE II | baseline
  Compare between APACHE II and AST/ALT ratio sensitivity as prognostic factors in patients with sepsis and septic shock.

IPD SHARING:
Plan to Share IPD: Undecided